CLINICAL TRIAL: NCT01483820
Title: A Phase I/II Trial of TPI-287 in Patients With Refractory or Recurrent Neuroblastoma and Medulloblastoma
Brief Title: Safety and Efficacy Study of TPI-287 in Neuroblastoma and Medulloblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Giselle Sholler (Other)
Collaborators: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Vice Study Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMTRC 004
Record Dates: First submitted 2011-11-28; First posted 2011-12-01 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma; Medulloblastoma
MeSH Terms: conditions — Neuroblastoma; Medulloblastoma | interventions — TPI-287

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TPI 287 (Experimental): Subjects will receive six cycles of intravenous (IV) TPI 287 at a dose of 125 mg/m2 on Days 1, 8 and 15 of a 21-day cycle.
  Interventions: Drug: TPI 287

INTERVENTIONS:
Drug: TPI 287 — Subjects will receive six cycles of intravenous (IV) TPI 287 at a dose of 125 mg/m2 on Days 1, 8 and 15 of a 21-day cycle.

SUMMARY:
The purpose of this research study is to evaluate a new investigational drug (TPI 287) for neuroblastoma and medulloblastoma. An investigational drug is one that has not yet been approved by the Food and Drug Administration. This investigational drug is called TPI 287. This study will look at the tumor's response to the study drug, TPI 287, as well as the safety and tolerability of the drug.

TPI 287 was shown to be effective in stopping tumor growth and was also shown to be safe in three different animal species. TPI 287 has been tested in humans in four clinical trials, and approximately 100 subjects with various types of cancers have received the drug, including a pediatric population in our previous Phase I trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically proven neuroblastoma or medulloblastoma and confirmation of refractory or recurrent disease with histologic confirmation at diagnosis or at the time of recurrence/progression
* Subjects must be age >12 months and diagnosed before the age of 21
* Measurable disease, including at least one of the following:
* Measurable tumor >10mm by CT or MRI
* Positive bone marrow biopsy/aspirate.
* Positive MIBG
* Current disease state must be one for which there is currently no known curative therapy
* Lansky Play Score or Karnofsky scale must be more than 30
* Subjects without bone marrow metastases must have an ANC > 750/μl and platelet count >50,000/μl
* Adequate Renal Function Defined As
* Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 or
* A serum creatinine based on age/gender
* Adequate liver function must be demonstrated, defined as:
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age
* SGPT (ALT) < 10 x upper limit of normal (ULN) for age
* SGOT (AST) < 10x upper limit of normal (ULN) for age
* No other significant organ toxicity defined as > Grade 2 by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE V4.0- http://ctep.cancer.gov/forms/CTCAEv4.pdf)
* A negative urine pregnancy test is required for female participants of child bearing potential (≥13 years of age or after onset of menses)
* Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.
* Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines
* Subjects may have received microtubulin inhibitors during previous therapies.

Exclusion Criteria:

* Anti-cancer Agents: Subjects who are currently receiving other anticancer agents are not eligible. Subjects must have fully recovered from the effects of prior chemotherapy (hematological and bone marrow suppression effects), generally at least 3 weeks from the most recent administration (6 weeks for nitrosoureas).
* Subjects who have received any myeloablative therapy within the previous 2 months.
* Subjects receiving anti-tumor therapy for their disease or any investigational drug concurrently
* Subjects with serious infection or a life-threatening illness (unrelated to tumor) that is > Grade 2 (NCI CTCAE V4.0), or active, serious infections requiring parenteral antibiotic therapy.
* Subjects with any other medical condition, including malabsorption syndromes, mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the interpretation of the results or which would interfere with a patient's ability to sign or the legal guardian's ability to sign the informed consent, and patient's ability to cooperate and participate in the study
* Subjects with known hypersensitivity to any of the components of the drugs to be administered on study

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Parikh, MD, Study Chair — Connecticut Children's Hospital; Giselle Sholler, MD, Principal Investigator — Beat Childhood Cancer at Atrium Health
Locations (8):
- United States (8):
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Arnold Palmer Hospital for Children- MD Anderson, Orlando, Florida
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- See also: Beat Childhood Cancer Consortium — http://www.beatcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TPI 287
Started | 8
Completed | 0
Not Completed | 8
Not completed — Lack of Efficacy | 6
Not completed — Adverse Event | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | TPI 287
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Phase I portion of trial- To determine the safety and tolerability of TPI 287 as a single agent in pediatric and young adult patients with refractory or recurrent neuroblastoma or medulloblastoma. Adverse events collected from time of first dose to 30 days past last dose and until all related events resolved, average of one year.
Time Frame: length of study +30 days
Measure: Number; unit: participants
Arm/Group | TPI 287
Number analyzed (Participants) | 8
participants | 6

2. Secondary Outcome: Number of Participants With Overall Response Assessed Using RECIST Criteria
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | TPI 287
Number analyzed (Participants) | 6
participants | 0

3. Secondary Outcome: Number of Days Participants Experienced Progression Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 3 years
Measure: Number; unit: Days
Arm/Group | TPI 287
Number analyzed (Participants) | 6
Days | 46

4. Secondary Outcome: Median Overall Survival (OS) of Participants
Description: Overall Survival (OS) and clinical benefit (ORR + stable disease, SD)
Time Frame: 3 years
Population: Not evaluated due to early closure. Study data does not exist.
Arm/Group | TPI 287
Number analyzed (Participants) | 0

5. Secondary Outcome: Quality of Life of Children Receiving TPI287 Using PedsQL Questionnaires
Description: To evaluate the impact of QOL of children receiving TPI287 using PedsQL questionnaires
Time Frame: 3 years
Population: QOL's not collected due to early closure of study. Data not collected or analyzed threfore no data exists.
Arm/Group | TPI 287
Number analyzed (Participants) | 0

6. Secondary Outcome: To Evaluate the Drug Levels and Pharmacokinetics (PK) of TPI 287 From Blood Samples at Multiple Time Points Within the First 24 Hours on Study.
Description: To evaluate the pharmacokinetics (PK) of TPI 287 in the Phase I population of this trial.
Time Frame: 1 year
Population: PK's not run due to early closure of study. Data not collected or analyzed threfore no data exists.
Arm/Group | TPI 287
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From date of first dose of TPI 287 until 30 days past last dose. Related AE's collected until resolution.
Arm/Group | TPI 287
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPI 287 (N=8)
Seizure (Nervous system disorders) | 1 (1)
Progression of Disease resulting in Death (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPI 287 (N=8)
alanine aminotransferase (ALT) increase (Hepatobiliary disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Aspartate aminotransferase (AST) increase (Hepatobiliary disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
fatigue (General disorders) | 1 (1)
Hypoglycemia (Endocrine disorders) | 1 (2)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Infusion related reaction (General disorders) | 2 (2)
Lymphocytopenia (Blood and lymphatic system disorders) | 1 (5)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 2 (3)
Nervous system disorders (Nervous system disorders) | 1 (1) — Tingling

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less